CLINICAL TRIAL: NCT01211054
Title: Epidemiologic Analysis for the Prevalence of Chronic Airway Diseases in Old Population in Korea
Brief Title: Epidemiologic Analysis for the Prevalence of Chronic Airway Diseases in Old Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chonbuk National University (Other)
Responsible Party: Yong Chul Lee, Chonbuk National University Medical School
Other Study IDs: RCPD old PFT
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: General Population, Spirometric Data, Medical Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Aim: To evaluate the spirometric data and the prevalence of chronic airway disease in old population (> 60 yrs) in Korea.

List to do

1. History taking
2. physical examination
3. Routine blood test
4. All spirometric data
5. In subgroup: further evaluation of allergic airway disease

ELIGIBILITY:
Inclusion Criteria:

* > 60 yrs olds
* no known specific respiratory diseases

Exclusion Criteria:

* taking any medication for respiratory diseases
* History of diagnosis as a respiratory disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For old people aged 60 yrs or more, the investigators will analyze their respiratory symptoms, spirometric data, smoking history, and atopic history in Korea.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-07